CLINICAL TRIAL: NCT04416815
Title: Integrating Health Promotion With and for Older People - eHealth: a Randomised Controlled Trial, in the Context of Good Quality Local Health Care
Brief Title: Integrating Health Promotion With and for Older People - eHealth
Acronym: IHOPe
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Göteborg University (Other)
Collaborators: The Swedish Research Council (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: GoteborgU-GPCC-IHOPe
Record Dates: First submitted 2020-04-02; First posted 2020-06-04 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-03

CONDITIONS: Frailty; Old Age
Keywords: Person-centredness; Telemedicine; RCT; e-health; Process Evaluation; Health Economic Evaluation; Health Plan; Partnership; Frailty; Elderly; Person-centred care; Patient-centred care; Person-centered care; Patient-centered care; Integrated care; Health promotion; eHealth
MeSH Terms: conditions — Frailty

STUDY DESIGN:
Intervention Model Description: RCT: All older people who give consent for participation and who fulfill the inclusion criteria will be randomised. Randomisation will be conducted by research nurses. Participants will be randomly assigned to either control or intervention group with a 1:1 allocation as per a computer generated randomisation. The control group will receive usual care. The intervention group will receive person-centred care intervention during 6 month on top of usual care.
Masking Description: The nature of the intervention means that neither participants nor the health care professionals (HCP) in the IHOPe intervention can be blinded to allocation in the RCT.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual care (No Intervention): The participants allocated to the control group received no intervention. However, they could, on their own initiative, approach the usual range of community or health services (e.g., home help services, rehabilitation, or medical care).
- eHealth (Experimental): The intervention will be delivered for 6 months on top of usual care.
  Interventions: Other: Integrating Health promotion with and for Older People - eHealth

INTERVENTIONS:
Other: Integrating Health promotion with and for Older People - eHealth — The intervention will be delivered for 6 months on top of usual care. It will be provided by HCPs. If needed one home visit to install the digital platform will be conducted. A HCP will introduce how to use the digital platform and create a personal account. The intervention starts with a person-centred phone-call where a health plan is co-created and potential team members to support this are identified and invited. The health plan includes the older persons' goals, internal and external resources, and need of support from health and/or social-services. This plan will be the point of departure for the forthcoming dialogue. A digital platform will open up for extended and safe communication and visualize the health planning between the older person and team-members in different settings. The older person and the HCP and involved team members on the digital platform will regularly evaluate the health plan and commonly agreed goals.
  Arms: eHealth

SUMMARY:
The Integrating Health promotion with and for Older People eHealth (IHOPe) project is expected to contribute vital knowledge on how older peoples capabilities and societal resources can be used in a more efficient way to promote health, self-management and enhance teamwork in partnership.The aim is to describe and evaluate this person-centered e-support intervention that promotes a sustainable partnership between community-dwelling frail older people and health and social care professionals. A digital platform, co-created with users and designed to create inclusion of individuals who today are living in a digital alienation, will be used in the health planning. In IHOPe frail older people will be able to identify their potential health issues but also their resources together with team partners from health- and social care, family or societal representatives. The intervention consists of person-centered phone calls with a health care professional as well as access to a digital platform that is accessible to the old person and invited team-partners. The project includes a randomized controlled trial, a process evaluation and a health economic evaluation. People 75 years or older screened as frail will be included. Also, in the process evaluation team-partners using the digital platform will be included. Specifically, this project is expected to reduce hospitalizations, result in improved or retained self-efficacy whilst being cost effective. Additionally, the project is expected to enhance frail older peoples opportunities to participate as an equal partner in their contacts with health and social services.

DETAILED DESCRIPTION:
Background:

Healthcare systems worldwide are not equipped to accommodate for the growing population of older people. In Sweden alone the proportion of people aged 65 years and older is estimated to increase to 23% by 2030. Furthermore, the number of people aged over 80 years in 2017 exceeded 500 000 and is expected to increase by around 50% by 2027. People in this age group often have an increased risk for developing frailty, multi-morbidity and functional impairments. Thus, there is an urgent call for innovative approaches to both promote health and to design a sustainable healthcare system that is accessible, resource effective and enables health in frail older people. Person-centered care (PCC) and digital health services are considered keystones in such a healthcare system redesign, and may enable efficient and resource effective teamwork that strengthens a preventive approach and promotes older people's self-efficacy. Previous and ongoing studies show that PCC can be delivered at a distance, but needs to be further developed from a teamwork aspect. Therefore, the IHOPe project focuses on integrating health promotion with and for frail older people by working as a team via a digital platform. To the best of our knowledge, no previous research has investigated the effectiveness of initiating health planning with and for frail older people through a PCC telephone support and eHealth intervention where patients are able to create a personal team by inviting informal and formal carers from both health and social care services into their health team if needed.

The overall aim is to describe and evaluate a person-centered eHealth intervention that promotes a sustainable partnership between community-dwelling frail older people and health and social care professionals.

Design:

The IHOPe trial is designed as a randomized, controlled, trial with two parallel groups and a primary endpoint 6 month after inclusion. Randomization will be performed through computer generated lists with a 1:1 allocation. In addition, the IHOPe project includes a pilot and feasibility study, a health economic evaluation and a process evaluation. The project is a complex intervention and as such features a multitude of influencing factors. The study design was guided by the revised Medical Research Council's (MRC) framework for complex interventions. The IHOPe project consists of two phases:

Phase 1: Develop and test feasibility of a person-centered eHealth intervention and pilot the RCT design.

Phase 2: Evaluate the effects, describe the process and perform a health economic evaluation of the person-centered eHealth intervention.

Studysetting/Context:

The IHOPe project is conducted in a middle sized city in Sweden and targets community dwelling older people, their family and friends and professionals working in local social and health care services. The intervention is delivered in an eHealth context and is coordinated by designated research nurses.

In Sweden there is an ongoing redesign of health care services towards good quality local health care [nära vård], which aims to strengthen primary care services and self-care. Health care costs in medical care are mainly financed through taxes and municipalities are responsible for services for older persons according to assessed needs. There are a number of actors representing different organizations involved in health and social care targeting older people. In addition, to such municipal services there are also private health and social care providers. It is also common that older people are receiving support or help from significant others.

Participants and recruitment procedure:

Participants will be recruited from either an emergency department or a primary care center in the western region of Sweden. Potential participants will be screened against inclusion and exclusion criteria for eligibility. Frailty screening will be performed by research assistants employed in the project at the emergency department or a primary care center if possible or otherwise by phone. The FRESH screening tool will be used which includes four short questions. If the answer is yes on two or more of these four questions patients is applicable for inclusion in the study. A Study Information letter and invitation to participate will be sent to eligible patients. After informed consent participants will be randomized to the intervention- or the control group.

Study population:

The RCT, targets frail older people aged 75 years or older living in ordinary housing. The feasibility study and process evaluation also include significant others and carers that are invited to the IHOPe platform.

Control group/usual care:

The participants allocated to the control group received no intervention. However, they could, on their own initiative, approach the usual range of community or health services (e.g., home help services, rehabilitation, or medical care).

Intervention/The eHealth support:

The IHOPe intervention is provided in addition to usual care for six months. It comprises an agreed upon number of person-centered phone calls (stimulating narration) and co-creation of care through a digital platform. The intervention aims to initiate partnership-building and to promote older people to identify and use their own capabilities and resources such as strong will, social relations, etc. During the intervention goals will be formulated and set in partnership to promote self-efficacy and the ability to cope with frailty in daily life. The older person (at times in collaboration with significant others) will together with a dedicated health care professional (HCP) formulate a person-centered health plan, which is then uploaded to the IHOPe platform. The health plan will focus on the older persons' goals, resources and needs, and experienced need of support from health and/or social care as well as family and friends to reach the goals. Depending on agreements during the phone-call family and friends and additional health or social care professionals may be invited to teamwork on the IHOPe platform. The health plan will be the point of departure for the forthcoming dialogue. IHOPe is provided in an eHealth context by designated HCPs trained in delivering PCC at a distance. Throughout the study, the HCP and patient (and team) will communicate to regularly evaluate the health plan and any need to reformulate the goals. The intervention is provided at a distance. If needed one home visit to install the digital platform (via the participant's smart tablet, smartphone or computer) will be conducted. A health professional will introduce how to use the digital platform and create a personal account.

ELIGIBILITY:
Inclusion Criteria:

* National registration within the Västra Götalands region (VGR), community dwelling people (men and women) aged 75 and older living in ordinary housing, and screened as frail at a primary care center or the emergency department but not hospitalized.

Exclusion Criteria:

* In need of palliative care in the final stages of life, no registered address, participating in any other conflicting randomised study, or cognitive dysfunctional (not oriented to time, place and person).

Min Age: 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2021-01-25 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
A composite of changes in general self-efficacy and need for hospital care | Baseline, 3
  The primary outcome is a composite of changes in general self-efficacy and need for hospital care for unscheduled reasons. Each participant will be classified as improved, deteriorated or unchanged if at 3 months:
  * Deteriorated: the participant's self-efficacy has decreased by ≥ 5 units (the minimal change of clinical significance), or the participant has been admitted to hospital for unscheduled reasons two times or more.
  * Improved: general self-efficacy has increased by ≥ 5 units and the participant has been admitted to hospital no more than once.
  * Unchanged: Neither deteriorated nor improved. (Questionnaire and medical record)

SECONDARY OUTCOMES:
Health-related quality of life by EuroQol 5 dimensions health state questionnaire (EQ5D) | Baseline, 3, 6, 12 months
  EQ5D is a generic measure of health status consisting of five dimensions (mobility, self-care, usual activities, pain/discomfort, anxiety/depression), each with responses indicating three levels of severity (no problems/some or moderate problems/extreme problems), the EQ Visual Analogue scale (EQ-VAS); a standard vertical 20 cm visual analogue scale for recording an individual's rating of their current health-related quality of life state raging from 'the best health you can imagine' to 'the worst health you can imagine'. (Questionnaire)
General Self Efficacy | Baseline, 3, 6, 12 months
  General Self-Efficacy Scale (GSE scale) is a 10-item self-assessment questionnaire designed to measure a broad and stable sense of personal competence to deal effectively with a variety of stressful situations. Ratings are made on a 4-point scale (1 = not at all true, 2 = hardly true, 3 = moderately true, 4 = exactly true) and are summed to a total score ranging from 10 to 40, where higher scores indicate greater self-efficacy. (Questionnaire)
Hospitalization | Baseline, 3, 6, 12 months
  The number of un-planned hospitalization. (Questionnaire and medical record)
ICEpop CAPability measure for Older people (ICECAP-O) | Baseline, 3, 6, 12 months
  The ICECAP-O capability index estimate quality of life in a broader sense, including five attributes (attachment, role, enjoyment, security, and control), each with four levels of response. (Questionnaire)
A composite of changes in general self-efficacy and need for hospital care for unscheduled reasons | Baseline, 6, 12 months
  A composite of changes in general self-efficacy and need for hospital care for unscheduled reasons at 6 and 12 moths.
Change in daily activities based on the ADL-staircase | Baseline, 3, 6, 12 months
  Independence from, or dependence on, another person in daily activities will be assessed based the ADL-staircase. The ADL-staircase applies a cumulative scale of ten well-defined personal activities (P-ADLs: bathing, dressing, going to the toilet, transfer, continence and feeding) and instrumental activities (I-ADLs: cleaning, shopping, transportation and cooking). Dependence is defined as receiving personal or directive assistance from another person. Participants living with another person is assessed as "independent" if they are capable of performing the activity independently. (Questionnaire)
Societal costs | Baseline, 3, 6, 12 months
  Resource use included in the economic evaluation will include: healthcare use (Region Västra Götaland), drug use and social care (National Board of Health and Welfare), as well as costs for informal care and other costs to the individual and/or family and friends related to the treatment collected from patient questionnaires and diaries. Costs (both reimbursements and out of pocket costs) for prescribed medications will be obtained from the Swedish Prescribed Drug Register. Cost per patient for healthcare use will be obtained from the register, and in resource use not recorded costs will be derived using national statistics, as will costs for social care and other costs reported in questionnaires. Informal care costs will be viewed as directs costs, and thus valued at the average wage and social security contribution of employing a formal caregiver.
Incremental cost-effectiveness Ratio (ICER) | Baseline, 3, 6, 12 months
  The ICER will be calculated as the difference in costs, between groups, divided by the corresponding difference in quality-adjusted life years (QALY). For the main analysis, QALYs will be derived from the EQ-5D index using the Swedish experience-based value set and using an area-under-the-curve calculation. Sensitivity analyses will be conducted using a society-based value set and the economic evaluation will also be conducted using a corresponding method with ICECAP-O as the health outcome.(Questionnaire)
Change in number of fall | Baseline, 3, 6, 12 months
  Self-reported number of fall during the last three months (Questionnaire)

OTHER OUTCOMES:
Change in burden of medicines use in everyday life based on The Living with medicines questionnaire version 3 (LMQ-3) | Baseline, 3, 6, 12 months
  Participants self-rate the following domains (relationships with health professionals, practical difficulties, interference with daily life, lack of effectiveness, side effects, general concerns, cost, and lack of autonomy) on a 5-point Likert scale (strongly agree to strongly disagree).
Change in the participants' self-rated overall level of medicines burden | Baseline, 3, 6, 12 months
  Participants assess the overall level of medicines burden on a 10 cm visual analogue scale from 0 (no burden at all) to 10 (extremely burdensome).

CONTACTS AND LOCATIONS:
Locations (1):
- Arvid Wallgrensbacke 7, Gothenburg, Gothenburg, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fried LP, Ferrucci L, Darer J, Williamson JD, Anderson G. Untangling the concepts of disability, frailty, and comorbidity: implications for improved targeting and care. J Gerontol A Biol Sci Med Sci. 2004 Mar;59(3):255-63. doi: 10.1093/gerona/59.3.m255. PMID 15031310
- [Background] Social Board. Being able to follow the patient's path through care Ways to link care events in the patient care process (Att kunna följa patientens väg genom vården Sätt att koppla samman vårdhändelser i patientens vårdprocess) socialstyrelsen, Editor. 2019, www.Socialstyrelsen.se, februari 2019 Stockholm.
- [Background] McCormack B. A conceptual framework for person-centred practice with older people. Int J Nurs Pract. 2003 Jun;9(3):202-9. doi: 10.1046/j.1440-172x.2003.00423.x. PMID 12801252
- [Background] Bandura A. Self-efficacy: toward a unifying theory of behavioral change. Psychol Rev. 1977 Mar;84(2):191-215. doi: 10.1037//0033-295x.84.2.191. No abstract available. PMID 847061
- [Background] Fors A, Ulin K, Cliffordson C, Ekman I, Brink E. The Cardiac Self-Efficacy Scale, a useful tool with potential to evaluate person-centred care. Eur J Cardiovasc Nurs. 2015 Dec;14(6):536-43. doi: 10.1177/1474515114548622. Epub 2014 Aug 22. PMID 25149667
- [Background] Ekman I, Swedberg K, Taft C, Lindseth A, Norberg A, Brink E, Carlsson J, Dahlin-Ivanoff S, Johansson IL, Kjellgren K, Liden E, Ohlen J, Olsson LE, Rosen H, Rydmark M, Sunnerhagen KS. Person-centered care--ready for prime time. Eur J Cardiovasc Nurs. 2011 Dec;10(4):248-51. doi: 10.1016/j.ejcnurse.2011.06.008. Epub 2011 Jul 20. PMID 21764386
- [Background] May CR, Mair FS, Dowrick CF, Finch TL. Process evaluation for complex interventions in primary care: understanding trials using the normalization process model. BMC Fam Pract. 2007 Jul 24;8:42. doi: 10.1186/1471-2296-8-42. PMID 17650326
- [Background] Craig P, Dieppe P, Macintyre S, Michie S, Nazareth I, Petticrew M; Medical Research Council Guidance. Developing and evaluating complex interventions: the new Medical Research Council guidance. BMJ. 2008 Sep 29;337:a1655. doi: 10.1136/bmj.a1655. PMID 18824488
- [Background] Grewal I, Lewis J, Flynn T, Brown J, Bond J, Coast J. Developing attributes for a generic quality of life measure for older people: preferences or capabilities? Soc Sci Med. 2006 Apr;62(8):1891-901. doi: 10.1016/j.socscimed.2005.08.023. Epub 2005 Sep 15. PMID 16168542
- [Background] Schultz-Larsen K, Avlund K. Tiredness in daily activities: a subjective measure for the identification of frailty among non-disabled community-living older adults. Arch Gerontol Geriatr. 2007 Jan-Feb;44(1):83-93. doi: 10.1016/j.archger.2006.03.005. Epub 2006 Nov 13. PMID 17095107
- [Background] Brooks R. EuroQol: the current state of play. Health Policy. 1996 Jul;37(1):53-72. doi: 10.1016/0168-8510(96)00822-6. PMID 10158943
- [Background] Schwarzer, R, Jerusalem, M, Generalized Self-Efficacy scale. In: Weinman J, Wright S, & Johnston M, eds. Measures in health psychology: A user's portfolio Causal and control beliefs. Windsor, England. NFER-NELSON 1995. pp. 35-37.
- [Background] Horder H, Gustafsson, S, Rydberg T, Skoog I, Waern M. A Cross-Cultural Adaptation of the ICECAP-O: Test-Retest Reliability and Item Relevance in Swedish 70-Year-Olds. Societies 2016. 6(4): p. 30.
- [Background] Sonn U, Grimby G, Svanborg A. Activities of daily living studied longitudinally between 70 and 76 years of age. Disabil Rehabil. 1996 Feb;18(2):91-100. doi: 10.3109/09638289609166023. PMID 8869511
- [Background] Gustafsson S, Horder H, Hammar IO, Skoog I. Face and content validity and acceptability of the Swedish ICECAP-O capability measure: Cognitive interviews with 70-year-old persons. Health Psychol Res. 2018 May 8;6(1):6496. doi: 10.4081/hpr.2018.6496. eCollection 2018 May 8. PMID 30596153
- [Background] Åsberg-Hulter, K., ADL-trappan (ADL- Staircase). 1990, Lund: Studentlitteratur.
- [Background] Rockwood K, Song X, MacKnight C, Bergman H, Hogan DB, McDowell I, Mitnitski A. A global clinical measure of fitness and frailty in elderly people. CMAJ. 2005 Aug 30;173(5):489-95. doi: 10.1503/cmaj.050051. PMID 16129869
- [Background] Katusiime B, Corlett SA, Krska J. Development and validation of a revised instrument to measure burden of long-term medicines use: the Living with Medicines Questionnaire version 3. Patient Relat Outcome Meas. 2018 May 28;9:155-168. doi: 10.2147/PROM.S151143. eCollection 2018. PMID 29881317
- [Background] Ebrahimi Z, Barenfeld E, Gyllensten H, Olaya-Contreras P, Fors A, Fredholm E, Fuller JM, Godarzi M, Krantz B, Swedberg K, Ekman I. Integrating health promotion with and for older people - eHealth (IHOPe) - evaluating remote integrated person-centred care : Protocol of a randomised controlled trial with effectiveness, health economic, and process evaluation. BMC Geriatr. 2023 Mar 27;23(1):174. doi: 10.1186/s12877-023-03866-6. PMID 36973667
- [Derived] Ebrahimi Z, Olaya-Contreras P, Goudarzi M, Ekman I. Experiences of a remote, person-centred intervention in older persons living with frailty - a qualitative study. BMC Geriatr. 2025 Oct 15;25(1):779. doi: 10.1186/s12877-025-06509-0. PMID 41094400
- See also: Study Protocol — https://bmcgeriatr.biomedcentral.com/articles/10.1186/s12877-023-03866-6